Informed consent

The Official Title of the study:

A study of behavioural changes in long-term home oxygen therapy in elderly patients with chronic obstructive pulmonary disease combined with mild cognitive impairment

date of the document:

9 May 2022

NCT number:

NCT06852716

Informed consent

Dear Uncle/Aunt,

Hello! I am XXX from the Respiratory Department of a hospital in Xiamen. Now I am conducting a project entitled "Study on the impact of health education Program based on BCW Theory on the compliance of long-term home oxygen therapy in elderly patients with chronic obstructive pulmonary disease complicated with mild cognitive Impairment". The purpose of this study is to help you take the initiative to promote health through **BCW** theory guidance. To improve self- management ability of long-term home oxygen therapy in compliance and elderly COPD patients with MCI. This study will last for 3 months and you are invited to participate in this study. If you are willing to participate in this study, you will be assessed for cognitive function,

emotional state, social psychology, blood oxygen saturation, lung function, etc.

Special note: We guarantee that all the information you participate in the study is confidential, and this investigation will not cause any harm to you and your family. Therefore, the evaluation and examination are provided free of charge, and you are free to choose to participate in or decline the study, and you have the right to withdraw from

the study at anytime.

If you are aware of the above information, please sign the Informed Consent box.

Thankyou again for your support and cooperation!

Signature of the consenting party:

Notification time: Year month date

I have explained to the study participant and obtained his/her understanding of informed consent.

**Investigator Signature:** 

Signature date: Year month date